CLINICAL TRIAL: NCT07106944
Title: Extended Tricyle Project Indonesia for Extended-spectrum Beta-lactamase Positive Klebsiella Pneumoniae and Escherichia Coli
Acronym: E-Trike
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dr. Sulianti Saroso Hospital, Jakarta (Unknown); Universitas Indonesia, Cipto Mangunkusumo National General Hospital (Unknown); RSUP Persahabatan Hospital, Jakarta, Indonesia (Unknown); National Institute for Public Health and the Environment (RIVM) (Other Government); Utrecht University (Other)
Responsible Party: Principal Investigator, Juliëtte Severin, Associate professor, MD PhD, Erasmus Medical Center
Other Study IDs: E-Trike
Record Dates: First submitted 2025-07-03; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Carriage of ESBL-positive Escherichia Coli; Carriage of ESBL-positive Klebsiella Pneumoniae
Keywords: ESBL; carriage; Escherichia coli; Klebsiella pneumoniae; One Health
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Bacterial isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community pregnant women: Pregnant women who do antenatal visits in primary health care centre (Puskesmas) located around Cipto Mangunkusumo Hospital, Persahabatan Hospital and Sulianti Saroso Hospital; Puskesmas Johar Baru, Puskesmas Pulogadung, and Puskesmas Koja. After informed consent, a rectal swab and throat swab will be taken. Basic demographic data will be recorded.
  Interventions: Other: Community pregnant women: rectal and throat swab

INTERVENTIONS:
Other: Community pregnant women: rectal and throat swab — Community pregnant women: rectal and throat swab

SUMMARY:
In 2019, Indonesia's first WHO Tricycle Project revealed alarming rates of extended-spectrum beta-lactamase (ESBL)-producing Escherichia coli across various sectors. The study found ESBL-producing E. coli in 40% of pregnant women, 57.7% of E. coli-induced bloodstream infections, 67.1% of broiler chicken, and 12.8% of total E. coli in water samples. In the first National Action Plan on Antimicrobial Resistance from Indonesia, the reduction of ESBL was identified as a clear goal. In E-Trike, Tricycle will be repeated, using the same methodology, to determine if a reduction has been achieved. Additionally, ESBL-positive Klebsiella pneumoniae will be included, as important pathogen for humans.

DETAILED DESCRIPTION:
Antimicrobial resistance (AMR) is a global threat and is considered to be a silent pandemic. It is estimated that in 2021, over 4.71 million deaths were associated with AMR, with 1.14 million attributed to AMR. In 2020, the World Health Organization (WHO) Global Antimicrobial Resistance and Use Surveillance System (GLASS) reported the prevalence of cefotaxime-, ceftriaxone, and ceftazidime-resistant Klebsiella pneumoniae from bloodstream infections in South Asian region was 75.9%, 77.4%, 74.8%, respectively. Based on the report from the Indonesian Society for Clinical Microbiologists in 2023, the prevalence of third-generation cephalosporin-resistant Klebsiella pneumoniae in Indonesia was 57%, while third-generation cephalosporin-resistant E. coli was 68%.

The WHO has been at the forefront of AMR through its Global Surveillance extended-spectrum beta-lactamase (ESBL)-positive E. coli Tricycle Project, which employs a "One Health" approach. This innovative surveillance program aims to obtain a comprehensive picture of AMR in humans, animals, and the environment, particularly in countries with limited surveillance capabilities. Indonesia's first pilot Tricycle Project revealed alarming rates of ESBL-producing E. coli across various sectors. The study found ESBL-producing E. coli in 40% of pregnant women, 57.7% of E. coli-induced bloodstream infections, 67.1% of broiler chicken, and 12.8% of total E. coli in water samples. These findings underscore the worrisome pattern of AMR in Indonesia and highlight the urgent need for expanded surveillance and control strategies.

Klebsiella pneumoniae is the second most common Enterobacterales found in humans; its role in animals and the environment is less clear, even more in the Indonesian setting. A better understanding of the presence of this human pathogen in other domains is needed, so that effective intervention strategies on AMR for the Indonesian situation can be designed.

In E-Trike, the original WHO Tricycle protocol (which already includes sample size calculation) will be used, with three modifications:

1. ESBL-K. pneumoniae (ESBL-Kp) will be included for all samples. Additionally, from pregnant women, not only rectal samples will be taken, but also throat samples, as previously it was shown that 15% of adults carry Kp in their throat in Indonesia.
2. In addition to the MacConkey agar supplemented with cefotaxime, CHROMagar plates will be used.
3. The sampling period will only be 5 months, instead of the 10 months that was used in the 2019 Tricycle. However, both "wet" and "dry" months will be included.

Primary aims:

* To determine the prevalence of ESBL-producing E. coli (ESBL-Ec) in humans (hospital and community), the food chain (animals), and the environment.
* To determine the prevalence of ESBL-producing Klebsiella pneumoniae (ESBL-Kp) in humans (hospital and community), the food chain (animals), and the environment.

Secondary aims:

* To compare the yield of the ESBL Chromagar™ plate compared to the MacConkey agar plate supplemented with 4 mg/L cefotaxime.
* To assess the susceptibility of the ESBL-Ec and ESBL-Kp to carbapenem antibiotics and other relevant classes of antibiotic.
* To understand the resistance mechanisms of ESBL-Ec and ESBL-Kp isolates using genomic analysis.

Setting The study will be performed in Jakarta, Indonesia.

Surveillance in humans will include:

Community: rectal and throat carriage in pregnant women in 3 puskesmas. From Hospitals: bloodstream infections with E. coli and K. pneumoniae, Cipto Mangunkusumo Hospital and Persahabatan Hospital; isolates will be included

Surveillance in food chain will include:

Chicken caeca from the live bird open market and slaughterhouse in Jakarta

Surveillance in the environment will include:

River water upstream and downstream, animal slaughter wastewater, human communal wastewater

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at antenatal visits

Exclusion Criteria:

* no informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women at antenatal visits in 3 puskesmas (public health centers)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of pregnant women in the community in Jakarta that carry ESBL-positive E. coli / Klebsiella pneumoniae in their rectum or throat | July 2025-March 2026
Number of ESBL-positive E. coli/K. pneumoniae among all blood cultures taken / all E. coli/K. pneumoniae from blood cultures | July 2025 - March 2026
Prevalence of ESBL-Ec and ESBL-Kp in the food chain (chicken) in Jakarta, Indonesia | July 2025 - March 2026
Prevalence of ESBL-Ec and ESBL-Kp in the environment (water) in Jakarta, Indonesia | July 2025 - March 2026

SECONDARY OUTCOMES:
Number of ESBL-Ec and ESBL-Kp ("yield") found using the ESBL Chromagar™ plate compared to the MacConkey agar plate supplemented with 4 mg/L cefotaxime per human subject or chicken or environmental sample included. | July 2025-March 2026
Number of ESBL-Ec and ESBL-Kp found in the study with resistance to carbapenem antibiotics and other relevant classes of antibiotic. | July 2025 - March 2026
The prevalence of ESBL resistant genes among the ESBL-Ec and ESBL-Kp isolates found in the study based on genomic analysis. | July 2025-March 2026

IPD SHARING:
Plan to Share IPD: Undecided
Due to privacy rules, it will only be provided upon reasonable request and completely anonymized.

REFERENCES:
- [Background] Puspandari N, Sunarno S, Febrianti T, Febriyana D, Saraswati RD, Rooslamiati I, Amalia N, Nursofiah S, Hartoyo Y, Herna H, Mursinah M, Muna F, Aini N, Risniati Y, Dhewantara PW, Allamanda P, Wicaksana DN, Sukoco R, Efadeswarni, Nelwan EJ, Cahyarini, Haryanto B, Sihombing B, Soares Magalhaes RJ, Kakkar M, Setiawaty V, Matheu J. Extended spectrum beta-lactamase-producing Escherichia coli surveillance in the human, food chain, and environment sectors: Tricycle project (pilot) in Indonesia. One Health. 2021 Sep 23;13:100331. doi: 10.1016/j.onehlt.2021.100331. eCollection 2021 Dec. PMID 34632041
- See also: Tricycle protocol WHO — https://www.who.int/publications/i/item/9789240021402